CLINICAL TRIAL: NCT02424318
Title: Effect of Topiramate on Cerebrovascular Response to Photic Stimulation in Migraineurs
Brief Title: Topiramate and Cerebrovascular Response in Migraineurs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Hyunwoo Nam, SMG-SNU Boramae Medical Center, SMG-SNU Boramae Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-2008-71
Record Dates: First submitted 2015-04-15; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topiramate (Experimental): topiramate 25mg twice for 1 week -> topiramate 50mg twice for 7 weeks
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — topiramate 25mg twice 1 week -> topiramate 50mg twice 7 weeks

SUMMARY:
The purpose of this study is to evaluate the effect of topiramate on cerebrovascular reactivity and mean flow velocity to photic stimulation in migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 65 years
* newly-diagnosed patients with migraine without aura (International Headache Society classification)
* symptom frequency (at least 2 episodes of migraine attack/month)

Exclusion Criteria:

* prior use of preventive medication
* patients with cardiovascular risk factors (hypertension, diabetes, hyperlipidemia, smoking)
* patients who take antihypertensive agent or antidepressant
* patients who were pregnant, breast-feeding or actively smoking
* patients with neurological or cerebrovascular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the Cerebrovascular reactivity | between baseline and after 2-month treatment of topiramate
  Transcranial Doppler sonography (TCD) was performed twice in migraineurs before and after the topiramate treatment during their interictal period of headache.
  Measurements: the mean flow velocity (MFV) of the right middle cerebral artery (MCA) and the left posterior cerebral artery (PCA). After 1 minute of adaptation period to the darkness, flashlights of 10 Hz were presented using a light source of an electroencephalography machine (PS40/R-220, Grass Technologies, West Warwick, USA). Recordings were performed for 10 cycles, and each cycle consisted of 10-second stimulation-on and 10-second stimulation-off.
  Calculation: Cerebrovascular reactivity (CVR) CVR = Δ V/Vb or Δ V/(VbxΔT) Where Vb is the baseline MFV, Δ V/Vb is the percentage MFV increase (amplitude), ΔT is the time from the onset of the stimulation to the peak MFV, and Δ V/(VbxΔT) is the slope of the MFV increase.

SECONDARY OUTCOMES:
Comparison of the mean flow velocities in the middle and posterior cerebral artery | between baseline and after 2-month treatment of topiramate
  Measurements: Same as outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Hyunwoo Nam, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center